CLINICAL TRIAL: NCT00658970
Title: A Combined Rising Single-dose (RSD) and Rising Multiple-dose (RMD)Phase 1 Study to Evaluate Safety, Tolerability and Pharmacokinetics of KX2-391 in Patients With Advanced Malignancies That Are Refractory to Conventional Therapies
Brief Title: Evaluation of KX2-391 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Allen Barnett/Chief Executivew Officer, Kinex Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KX01-01-07
Record Dates: First submitted 2008-01-15; First posted 2008-04-16 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Solid Tumors; Lymphoma
Keywords: Open label; Dose escalation
MeSH Terms: conditions — Lymphoma | interventions — tirbanibulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: KX2-391 — 2 mg (starting dose)rising dose, oral dosing, twice daily, 21 day cycle(s); until progression or unacceptable toxicity develops

SUMMARY:
The purpose of this Phase 1 study is to determine the safety and tolerability of KX2-391 in cancer patients.

DETAILED DESCRIPTION:
The purpose of this first in human study is to determine the safety and pharmacokinetics of KX2-391 in patients with solid tumors and lymphoma, who are refractory to conventional cancer treatments. In addition, pharmacodynamics will be evaluated using biomarkers in peripheral blood mononuclear cells and in tissue biopsy samples.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Adults over age 18 years of age
* Confirmed advanced solid tumor or lymphoma that may be metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; patients with treated brain or ocular metastases are also eligible
* ECOG performance status of 0-2
* Life expectancy of at least 14 weeks
* Adequate bone marrow reserve
* Adequate liver function as demonstrated by serum bilirubin, alanine aminotransferase (ALT), aspartate transaminase (AST) and alkaline phosphatase (ALP)
* Adequate renal function (serum creatinine </= 1.5 x ULN or calculated creatinine clearance > 60 ml/min)
* Normal coagulation profile (PT/INR and aPTT within institutional normal limits) for those who give consent to tumor biopsy, within 1 week prior to the procedure.
* Negative pregnancy test for females at Screening, preferably done within 1 week before Day 1 of dosing (not applicable to patients with bilateral oophorectomy and/or hysterectomy)
* Willing to abstain from sexual activity or practice physical barrier contraception 28 days before Day 1 of dosing and 6 months after the last dose for the patient
* Signed written informed consent for tumor biopsy for the additional 10 subjects that will be dosed at the MTD and who have accessible tumors

Exclusion Criteria:

* Unresolved toxicity of higher than Grade 1 severity from previous anti-cancer treatment or investigational agents
* Receiving or having received investigational agents or systemic anti-cancer agents within 14 days of Day 1 of dosing or 28 days for those agents with unknown elimination half-lives or half-lives of greater than 50 hours
* Received extensive radiation therapy including sternum, pelvis, scapulae, vertebrae or skull, </= 4 weeks or low dose palliative radiation therapy limited to limbs </= 1 week prior to starting study drug, or who have not recovered from side effects of such therapy
* Currently taking hormones (i.e., estrogen contraceptives, hormone replacement, anti-estrogen), anti-platelet agents or anti-coagulants, e.g. coumadin, except for those who are on prophylactic doses of anti-coagulants for indwelling venous catheters
* Use of strong inhibitors or inducers of cytochrome P450 3A4 enzymes 2 weeks or 5 half-lives prior to Day 1 of dosing and during the study (refer to Appendix 3)
* Pregnant or breast-feeding
* Major surgery within 4 weeks prior to Day 1 of dosing
* Major surgery to the upper gastrointestinal tract, or inflammatory bowel disease, malabsorption syndrome or other medical condition that may interfere with oral absorption
* Signs or symptoms of end organ failure, major chronic illnesses other than cancer, or any severe concomitant conditions which, in the opinion of the investigator, makes it undesirable for the subject to participate in the study or which could jeopardize compliance with the protocol
* History of angina pectoris, coronary artery disease or cerebrovascular accident, transient ischemic attack or cardiac arrhythmia requiring medical therapy
* Evidence of hepatitis B or C, human immunodeficiency (HIV) infection, coagulation disorders, or hemolytic conditions, e.g. sickle cell anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose of the drug | 64 days

SECONDARY OUTCOMES:
Pharmacokinetics, Pharmacodynamics, Efficacy | 64 days

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, M.D., Principal Investigator — M.D. Anderson Cancer Center; Roger B Cohen, M.D., Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas